CLINICAL TRIAL: NCT03345472
Title: Vectors Post Market: A Study to Assess Pain Relief Using Spinal Cord Stimulation (SCS) With High Dose (HD) Stimulation Parameters
Brief Title: Vectors Post Market: A Study to Assess Pain Relief Using Spinal Cord Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT17053
Record Dates: First submitted 2017-11-14; First posted 2017-11-17 (Actual); Results first posted 2020-03-20 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treated (Experimental): Enrolled subjects who are implanted with a spinal cord stimulation system that is activated.
  Interventions: Device: Spinal Cord Stimulation System

INTERVENTIONS:
Device: Spinal Cord Stimulation System — Implanted neurostimulation system (neurostimulator and leads) with high dose stimulation parameters.
  Other Names: Medtronic RestoreSensor SureScan MRI neurostimulation system; Medtronic Intellis AdaptiveStim neurostimulation system

SUMMARY:
This is a prospective, single-arm, multi-center study evaluating the efficacy of spinal cord stimulation (SCS) therapy for pain relief using high dose (HD) stimulation parameters delivered to neural targets identified during current commercial trial stimulation procedures. The study will evaluate changes in back and leg pain from baseline to 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Candidate per labeling for an SCS system as an aid in the management of chronic, intractable low back and leg pain
* Presence of low back and leg pain
* Moderate to crippled disability due to pain
* Stable pain medications for back and leg pain for at least 28 days prior to enrollment
* Willing and able to not increase pain medications through the 3-Month visit

Exclusion Criteria:

* Previously trialed or implanted with stimulator or intrathecal drug delivery system
* Current diagnosis of moderate to severe central lumbar spinal stenosis
* Major psychiatric comorbidity or other progressive diseases
* Serious drug-related behavioral issues
* Pregnant or planning on becoming pregnant
* Unable to achieve supine position

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2019-02-04 (Actual); Study Completion 2019-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vectors Post Market Clinical Research Study Team, Study Director — Medtronic Restorative Therapies, Pain Therapy
Locations (20):
- United States (20):
  - Pain Consultants of San Diego, La Mesa, California
  - Restore Orthopedics and Spine Center, Orange, California
  - Center for Interventional Pain and Spine, Wilmington, Delaware
  - Pain Care, Stockbridge, Georgia
  - National Spine and Pain, Oxon Hill, Maryland
  - Michigan Pain Consultants, Wyoming, Michigan
  - Comprehensive and Interventional Pain Management, Henderson, Nevada
  - The Pain Management Center, Voorhees Township, New Jersey
  - University of Rochester Neurosurgery Partners Pain Management, Rochester, New York
  - Carolinas Pain Center, Huntersville, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Lehigh Valley Healthcare Network, Allentown, Pennsylvania
  - Saint Luke's Neurosurgical Associates, Bethlehem, Pennsylvania
  - Pain Diagnostics and Interventional Care, Sewickley, Pennsylvania
  - Delaware Valley Pain and Spine Institute, Trevose, Pennsylvania
  - Lowcountry Orthopaedics/Coastal Carolina Research Center, Charleston, South Carolina
  - Carolina Center for Advanced Management of Pain, Spartanburg, South Carolina
  - Precision Spine Care, Tyler, Texas
  - Carilion Clinic Roanoke Memorial Hospital, Roanoke, Virginia
  - Northwest Pain Care, Spokane, Washington

REFERENCES:
- [Derived] Hatheway JA, Mangal V, Fishman MA, Kim P, Shah B, Vogel R, Galan V, Severyn S, Weaver TE, Provenzano DA, Chang E, Verdolin MH, Howes G, Villarreal A, Falowski S, Hendrickson K, Stromberg K, Davies L, Johanek L, Kelly MT. Long-Term Efficacy of a Novel Spinal Cord Stimulation Clinical Workflow Using Kilohertz Stimulation: Twelve-Month Results From the Vectors Study. Neuromodulation. 2021 Apr;24(3):556-565. doi: 10.1111/ner.13324. Epub 2020 Dec 9. PMID 33296127

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 175 subjects were enrolled. 32 exited before the spinal cord stimulation trial. 143 subjects started the trial and 12 exited during the trial. 131 subjects completed the trial: 117 had a successful high dose (HD) trial; the 14 with unsuccessful HD trial were exited. Of the 117, 14 exited before implant and 103 were implanted (Treated Arm).
Period: Implant to 3 Months
Arm/Group | Treated
Started | 103
Completed | 99
Not Completed | 4
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 1
Not completed — Adverse Event | 1
Period: 3 Months to 12 Months
Arm/Group | Treated
Started | 99
Completed | 91
Not Completed | 8
Not completed — Physician Decision | 3
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treated
Number analyzed (Participants) | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 93
  Unknown or Not Reported | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 92
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 103
Years from pain onset to enrollment [Mean (Standard Deviation); unit: years] | 12.9 (11.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Overall Pain Intensity on the Visual Analog Scale (0-100)
Description: Demonstrate a significant improvement in overall pain intensity as measured by the Visual Analog Scale (VAS).
  The VAS ranges from 0 (no pain) to 100 (worst pain imaginable). The change in overall pain intensity is calculated as the Baseline VAS minus the 3-month VAS, where a positive value indicates an improvement (ie, reduction) in pain from Baseline to 3 months. Higher values represent a larger reduction (ie, greater improvement) in pain.
  The change in overall pain intensity as measured by the VAS can range from -100 (worsening in pain from 0 at baseline to 100 at 3 months) to 100 (improvement in pain from 100 at baseline to 0 at 3 months). It should be noted that while the change in VAS can range from -100 to 100, no subjects had a VAS of 0 at baseline, as the presence of pain was required for eligibility for inclusion in the study.
Time Frame: Baseline to 3 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Treated
Number analyzed (Participants) | 103
units on a scale | 45.4 (2.6)

2. Secondary Outcome: Overall Pain Efficacy Responder Rate
Description: Characterize the overall pain efficacy responder rate, where the responder rate is the percentage of subjects who experience at least a 50% improvement in overall pain, as measured by the Visual Analog Scale (VAS).
  The VAS ranges from 0 (no pain) to 100 (worst pain imaginable). The percent improvement for each subject was calculated as [100*(Baseline VAS - 3-month VAS)/Baseline VAS], where a positive number represents an improvement, and the larger the number the greater the percent improvement. If the percent improvement from baseline to 3 months was at least 50%, the subject was considered a responder.
  The percentage of subjects who experience at least a 50% improvement in overall pain can range from 0% (no responders) to 100% (all responders).
Time Frame: Baseline to 3 months
Measure: Number (95% Confidence Interval); unit: percent of subjects who are responder
Arm/Group | Treated
Number analyzed (Participants) | 103
percent of subjects who are responder | 68.3 [59.0 to 77.5]

3. Secondary Outcome: Low Back Pain Efficacy Responder Rate
Description: Characterize the low back pain efficacy responder rate, where the responder rate is the percentage of subjects who experience at least a 50% improvement in low back pain, as measured by the Visual Analog Scale (VAS).
  The VAS ranges from 0 (no pain) to 100 (worst pain imaginable). The percent improvement for each subject was calculated as [100*(Baseline VAS - 3-month VAS)/Baseline VAS], where a positive number represents an improvement, and the larger the number the greater the percent improvement. If the percent improvement from baseline to 3 months was at least 50%, the subject was considered a responder.
  The percentage of subjects who experience at least a 50% improvement in low back pain can range from 0% (no responders) to 100% (all responders).
Time Frame: Baseline to 3 months
Measure: Number (95% Confidence Interval); unit: percent of subjects who are responders
Arm/Group | Treated
Number analyzed (Participants) | 103
percent of subjects who are responders | 59.8 [49.9 to 69.7]

4. Secondary Outcome: Leg Pain Efficacy Responder Rate
Description: Characterize the leg pain efficacy responder rate, where the responder rate is the percentage of subjects who experience at least a 50% improvement in leg pain, as measured by the Visual Analog Scale (VAS).
  The VAS ranges from 0 (no pain) to 100 (worst pain imaginable). The percent improvement for each subject was calculated as [100*(Baseline VAS - 3-month VAS)/Baseline VAS], where a positive number represents an improvement, and the larger the number the greater the percent improvement. If the percent improvement from baseline to 3 months was at least 50%, the subject was considered a responder.
  The percentage of subjects who experience at least a 50% improvement in leg pain can range from 0% (no responders) to 100% (all responders).
Time Frame: Baseline to 3 months
Measure: Number (95% Confidence Interval); unit: percent of subjects who are responders
Arm/Group | Treated
Number analyzed (Participants) | 103
percent of subjects who are responders | 77.4 [69.1 to 85.7]

ADVERSE EVENTS:
Time Frame: 12 months post-device activation
Description: Adverse events related to the implanted spinal cord stimulation system, accessories, surgical procedures, and therapy were collected.
  The sum of subjects affected within each individual event may not add to the total number of subjects affected, as subjects may have experienced more than 1 type of event.
Arm/Group | Treated
All-Cause Mortality (participants affected / at risk) | 1/103
Serious Adverse Events (participants affected / at risk) | 1/103
Other Adverse Events (participants affected / at risk) | 36/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treated (N=103)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treated (N=103)
Paraesthesia (Nervous system disorders) | 19 (25)
Device stimulation issue (Product Issues) | 11 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Per the Clinical Investigation Plan, all proposed publications must be reviewed and approved by Medtronic prior to publication.

DOCUMENTS (2):
  • Study Protocol (2018-05-08): https://cdn.clinicaltrials.gov/large-docs/72/NCT03345472/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-21): https://cdn.clinicaltrials.gov/large-docs/72/NCT03345472/SAP_001.pdf